CLINICAL TRIAL: NCT04872738
Title: Patient Experiences With the COVID-19 Vaccination After Breast Cancer Treatment
Acronym: LymphVAX
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Alphonse Taghian, Director, Lymphedema Research Program, Massachusetts General Hospital
Other Study IDs: 21-528
Record Dates: First submitted 2021-05-02; First posted 2021-05-04 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer Related Lymphedema; Covid19
Keywords: Breast Cancer; Vaccination; Lymphadenopathy
MeSH Terms: conditions — Breast Cancer Lymphedema; COVID-19; Breast Neoplasms; Lymphadenopathy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaccinated Breast Cancer Patients [mRNA vaccine - Moderna, Pfizer]: Patients who enroll in the trial and decided to get the COVID-19 vaccine will complete surveys to indicate their experiences, side effects, location of vaccination (i.e. right arm, left arm, or leg). This information will be analyzed in conjunction with their breast cancer treatment history and lymphedema measurements.
  Participants were separated into two different cohorts for analysis, Cohort 1 being those who received an mRNA vaccine for their primary vaccination series (two doses of Moderna or Pfizer) and Cohort 2 being those who received a non-mRNA vaccination for their primary vaccination series (one dose of Johnson & Johnson).
  Interventions: Other: Survey
- Vaccinated Breast Cancer Patients [non-mRNA vaccine - Johnson & Johnson]: Patients who enroll in the trial and decided to get the COVID-19 vaccine will complete surveys to indicate their experiences, side effects, location of vaccination (i.e. right arm, left arm, or leg). This information will be analyzed in conjunction with their breast cancer treatment history and lymphedema measurements.
  Participants were separated into two different cohorts for analysis, Cohort 1 being those who received an mRNA vaccine for their primary vaccination series (two doses of Moderna or Pfizer) and Cohort 2 being those who received a non-mRNA vaccination for their primary vaccination series (one dose of Johnson & Johnson).
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Patients in all groups will complete surveys about their experience with the vaccination and any side effects they may have experienced.

SUMMARY:
This study aims to elicit patient experiences, choices, and side effects associated with the COVID-19 vaccine after breast cancer surgery. Lymph node swelling is a known and common side effect of both the Moderna and Pfizer COVID-19 vaccines. This is the body's normal reaction to the vaccine. It is worrisome that lymph node swelling after the vaccine mimics that found in breast cancer which has spread to the lymph nodes. This side effect will cause worry and anxiety amongst patients as a result. For patients who have had lymph node removal (axillary lymph node dissection or sentinel lymph node biopsy) and are at risk of lymphedema, the investigators are concerned that the lymph node swelling may tax the lymphatic system and incite lymphedema in those at risk or worsen it in those with BCRL. Fear of lymphedema is high in this population and the investigators need to better understand what risk, if any, lymph node swelling after the COVID-19 vaccine imparts to BCRL risk.

DETAILED DESCRIPTION:
* Hypothesis 1: Patients will choose to receive the vaccine on the arm contralateral to axillary lymph node removal, or in the lower extremity if they have had bilateral axillary lymph node removal
* Hypothesis 2: Patients with a history of breast cancer will experience axillary lymph node swelling after receiving the COVID-19 vaccine at the same rate as the general population
* Hypothesis 3: Patients with axillary surgery who develop lymph nodes swelling in the ipsilateral side might be at increased risk of developing lymphedema

ELIGIBILITY:
Inclusion Criteria:

* Female patients who are
* ≥18 years of age and have a
* History of breast cancer For the MGH site, patients must have
* Received some breast cancer treatment at MGH or its affiliates
* Received perometry measurements to measure arm volume at MGH

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with a history of breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 714 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alphonse G Taghian, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Juhel BC, Brunelle CL, Bernstein MC, Smith LH, Jung AW, Ababneh HS, Hausman EK, Bucci LK, Bernstein T, Naoum GE, Taghian AG. Side effects of COVID-19 vaccinations in patients treated for breast cancer. Clin Exp Med. 2023 Nov;23(7):3671-3680. doi: 10.1007/s10238-023-01050-z. Epub 2023 Apr 8. PMID 37031282

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We excluded 44 incomplete surveys or surveys from patients who received the first vaccine prior to breast cancer treatment, resulting in data from 670 patients for analysis.
Period: Dose 1/Primary Series Survey
Arm/Group | Vaccinated Breast Cancer Patients [mRNA Vaccine - Moderna, Pfizer] | Vaccinated Breast Cancer Patients [Non-mRNA Vaccine - Johnson & Johnson]
Started | 621 | 49
Completed | 621 | 49
Not Completed | 0 | 0
Period: Booster Survey
Arm/Group | Vaccinated Breast Cancer Patients [mRNA Vaccine - Moderna, Pfizer] | Vaccinated Breast Cancer Patients [Non-mRNA Vaccine - Johnson & Johnson]
Started (Only, and all, participants from the 'Dose 1/Primary Series Survey' period were sent the Booster Survey for completion. The participants who chose to complete the Booster Survey were then included in the 'Booster Survey' period.) | 621 | 49
Completed | 469 | 34
Not Completed | 152 | 15
Not completed — Did not respond or did not receive booster dose at the time of survey distribution | 152 | 15

BASELINE CHARACTERISTICS:
Population: Demographic and breast cancer-related characteristics for the 621 patients receiving an mRNA primary vaccine series and the 49 patients receiving a non-mRNA primary vaccine series were presented.
Groups:
- Vaccinated Breast Cancer Patients [mRNA Vaccine - Moderna, Pfizer]: Patients who enroll in the trial and decided to get the COVID-19 vaccine will complete surveys to indicate their experiences, side effects, location of vaccination (i.e. right arm, left arm, or leg). This information will be analyzed in conjunction with their breast cancer treatment history and lymphedema measurements.
  Participants were separated into two different cohorts for analysis, Cohort 1 being those who received an mRNA vaccine (Moderna, Pfizer) and Cohort 2 being those who received a non-mRNA vaccination (Johnson & Johnson). Demographic data for Cohort 2 is not included, as this cohort was not included in the primary analysis and therefore its data was not pulled.
- Total: Total of all reporting groups
Arm/Group | Vaccinated Breast Cancer Patients [mRNA Vaccine - Moderna, Pfizer] | Vaccinated Breast Cancer Patients [Non-mRNA Vaccine - Johnson & Johnson] | Total
Number analyzed (Participants) | 621 | 49 | 670
Age, Continuous [Median (Full Range); unit: years] | 53 [26.2 to 83.6] | 53.8 [31.2 to 74.4] | 53.1 [26.2 to 83.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 621 | 49 | 670
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI, Continuous [Median (Full Range); unit: kg/m²] — Population: There was missing data for 2 participants in regards to BMI for the mRNA vaccine cohort and missing data for 3 participants in regards to BMI for the non-mRNA vaccine cohort.
  kg/m²
    number analyzed (Participants) | 619 | 46 | 665
    (all) | 26.0 [15.8 to 50.4] | 27.2 [19.2 to 47.3] | 26.0 [15.8 to 50.4]
BMI > 25 [Count of Participants; unit: Participants] — Population: There was missing data for 2 participants in regards to BMI for the mRNA vaccine cohort and missing data for 3 participants in regards to BMI for the non-mRNA vaccine cohort.
  Participants
    number analyzed (Participants) | 619 | 46 | 665
    (all) | 356 | 27 | 383
Mastectomy with Reconstruction [Count of Participants; unit: Participants] | 222 | 11 | 233
Mastectomy without Reconstruction [Count of Participants; unit: Participants] | 51 | 6 | 57
Lumpectomy [Count of Participants; unit: Participants] | 348 | 31 | 379
Axillary Lymph Node Dissection [Count of Participants; unit: Participants] | 176 | 18 | 194
Sentinel Lymph Node Biopsy [Count of Participants; unit: Participants] | 393 | 24 | 417
No Nodal Surgery [Count of Participants; unit: Participants] | 52 | 7 | 59
Regional Lymph Node Radiation [Count of Participants; unit: Participants] | 188 | 20 | 208
Neoadjuvant +/- adjuvant chemotherapy [Count of Participants; unit: Participants] | 109 | 11 | 120
Adjuvant chemotherapy, only [Count of Participants; unit: Participants] | 196 | 14 | 210
Time between breast surgery and first dose [Median (Full Range); unit: months] — Population: There was missing data for 3 participants in regards to date of surgery for the non-mRNA vaccine cohort.
  months
    number analyzed (Participants) | 621 | 46 | 667
    (all) | 69.0 [0.13 to 361.5] | 85.4 [3.0 to 350.4] | 70.1 [0.13 to 361.5]

OUTCOME MEASURES:

1. Primary Outcome: COVID-19 Vaccination on Contralateral vs Ipsilateral Arm
Description: The investigators expect 90% of participants to receive the COVID-19 vaccine on their contralateral (unaffected) arm.
  This outcome measure is looking at the number of participants who received the COVID-19 vaccine on the side of breast cancer treatment vs those who received the vaccine on the opposite side of breast cancer treatment.
  Patients with bilateral cancer were excluded from this analysis due to the nature of breast cancer laterality categorization.
Time Frame: This was a survey study of patients with breast surgery for breast cancer. Participants replied to the online survey up to 361.5 months post their breast surgery (median 69.0 months). This was the study's reported timeframe in the published manuscript.
Population: The cohort of patients who received a non-mRNA vaccine was not included in the analysis, as only a small proportion of the population received this vaccine type. Consequently, data on this group were not collected.
Measure: Count of Participants; unit: Participants
Groups:
- Vaccinated Breast Cancer Patients Dose 1 [mRNA vaccine - Moderna, Pfizer]; Vaccinated Breast Cancer Patients Dose 2 [mRNA vaccine - Moderna, Pfizer]; Vaccinated Breast Cancer Patients Booster [mRNA vaccine - Moderna, Pfizer]; Vaccinated Breast Cancer Patients [non-mRNA vaccine - Johnson & Johnson]: Patients who enroll in the trial and decided to get the COVID-19 vaccine will complete surveys to indicate their experiences, side effects, location of vaccination (i.e. right arm, left arm, or leg). This information will be analyzed in conjunction with their breast cancer treatment history and lymphedema measurements.
  Participants were separated into two different cohorts for analysis, Cohort 1 being those who received an mRNA vaccine for their primary vaccination series (two doses of Moderna or Pfizer) and Cohort 2 being those who received a non-mRNA vaccination for their primary vaccination series (one dose of Johnson & Johnson).
Arm/Group | Vaccinated Breast Cancer Patients Dose 1 [mRNA vaccine - Moderna, Pfizer] | Vaccinated Breast Cancer Patients Dose 2 [mRNA vaccine - Moderna, Pfizer] | Vaccinated Breast Cancer Patients Booster [mRNA vaccine - Moderna, Pfizer] | Vaccinated Breast Cancer Patients [non-mRNA vaccine - Johnson & Johnson]
Number analyzed (Participants) | 554 | 554 | 405 | 0
Participants
  Patients who received the vaccine contralateral to breast cancer treatment | 432 | 435 | 331 |
  Patients who received the vaccine ipsilateral to breast cancer treatment | 122 | 119 | 74 |

2. Primary Outcome: Lymph Node (LN) Swelling After COVID-19 Vaccine
Description: The investigators expect 10-15% of participants to experience lymph node swelling after receiving the Pfizer or Moderna vaccines.
  The outcome measure analyzes the number of participants who experienced LN swelling after receiving each dose of their COVID-19 vaccines. The analysis looked at what location on the body lymph node swelling occurred (axilla vs supraclavicular region), which side of the body this swelling occurred in relation to the side of the body that received the vaccine (ipsilateral vs contralateral), and which side of the body this swelling occurred in relation to the side of the body the patient has/had breast cancer (ipsilateral vs contralateral).
  Patients with bilateral cancer were excluded from the analysis of LN swelling in relation to both the vaccine and breast cancer laterality due to the nature of BC laterality categorization.
  Analysis on breast cancer laterality and LN swelling was not conducted for the non-mRNA vaccine (Johnson & Johnson) group.
Time Frame: as for outcome 1
Population: The first row, 'Lymph node (LN) swelling, general', reports the number of subjects who reported LN swelling. We then analyzed, of the subjects who indicated that they experienced LN swelling, the laterality in which this swelling occurred. These data are represented in rows 2 through 5.
  In the analysis of LN swelling laterality related to both vaccine and BC laterality, the population size was the number of participants vaccinated on the specified side (only conducted for mRNA vaccines).
Measure: Count of Participants; unit: Participants
Groups:
- Vaccinated Breast Cancer Patients Dose 1 [non-mRNA vaccine - Johnson & Johnson]; Vaccinated Breast Cancer Patients Booster [non-mRNA vaccine - Johnson & Johnson]: Patients who enroll in the trial and decided to get the COVID-19 vaccine will complete surveys to indicate their experiences, side effects, location of vaccination (i.e. right arm, left arm, or leg). This information will be analyzed in conjunction with their breast cancer treatment history and lymphedema measurements.
  Participants were separated into two different cohorts for analysis, Cohort 1 being those who received an mRNA vaccine for their primary vaccination series (two doses of Moderna or Pfizer) and Cohort 2 being those who received a non-mRNA vaccination for their primary vaccination series (one dose of Johnson & Johnson).
Arm/Group | Vaccinated Breast Cancer Patients Dose 1 [mRNA vaccine - Moderna, Pfizer] | Vaccinated Breast Cancer Patients Dose 2 [mRNA vaccine - Moderna, Pfizer] | Vaccinated Breast Cancer Patients Booster [mRNA vaccine - Moderna, Pfizer] | Vaccinated Breast Cancer Patients Dose 1 [non-mRNA vaccine - Johnson & Johnson] | Vaccinated Breast Cancer Patients Booster [non-mRNA vaccine - Johnson & Johnson]
Number analyzed (Participants) | 621 | 621 | 469 | 49 | 34
Participants
  Lymph node (LN) swelling, general | 61 | 80 | 53 | 4 | 1
  LN swelling: Supraclavicular, Contralateral to Vaccine: number analyzed (Participants) | 61 | 80 | 53 | 49 | 34
  LN swelling: Supraclavicular, Contralateral to Vaccine | 11 | 16 | 5 | 0 | 0
  LN swelling: Supraclavicular, Ipsilateral to Vaccine: number analyzed (Participants) | 61 | 80 | 53 | 49 | 34
  LN swelling: Supraclavicular, Ipsilateral to Vaccine | 18 | 21 | 17 | 1 | 0
  LN swelling: Axillary, Contralateral to Vaccine: number analyzed (Participants) | 61 | 80 | 53 | 49 | 34
  LN swelling: Axillary, Contralateral to Vaccine | 28 | 36 | 13 | 0 | 1
  LN swelling: Axillary, Ipsilateral to Vaccine: number analyzed (Participants) | 61 | 80 | 53 | 49 | 34
  LN swelling: Axillary, Ipsilateral to Vaccine | 33 | 50 | 38 | 3 | 0
  LN swelling ipsilateral to vaccine, contralat. to BC (among pts who received dose contralat. to BC): number analyzed (Participants) | 432 | 435 | 331 | 0 | 0
  LN swelling ipsilateral to vaccine, contralat. to BC (among pts who received dose contralat. to BC) | 33 | 48 | 40 |  |
  LN swelling contralat. to vaccine, ipsilateral to BC (among pts who received dose contralat. to BC): number analyzed (Participants) | 432 | 435 | 331 | 0 | 0
  LN swelling contralat. to vaccine, ipsilateral to BC (among pts who received dose contralat. to BC) | 30 | 42 | 12 |  |
  Ipsilateral to vaccine and to BC (among pts who received dose ipsilateral to BC): number analyzed (Participants) | 122 | 119 | 74 | 0 | 0
  Ipsilateral to vaccine and to BC (among pts who received dose ipsilateral to BC) | 14 | 17 | 10 |  |
  Contralateral to vaccine and to BC (among pts who received dose ipsilateral to BC): number analyzed (Participants) | 122 | 119 | 74 | 0 | 0
  Contralateral to vaccine and to BC (among pts who received dose ipsilateral to BC) | 6 | 7 | 5 |  |

3. Primary Outcome: Duration of Lymph Node Swelling as a Side Effect of mRNA and Non-mRNA Vaccines
Description: The outcome measure will be analyzing the reported duration of lymph node swelling, categorized by the location at which lymph node swelling occurred (the axilla vs supraclavicular region) and which side of the body this swelling occurred in relation to the side of the body that received the vaccine injection (ipsilateral vs contralateral). The main aim of this paper was to report the side effects of the mRNA COVID-19 vaccines in patients treated for breast cancer.
Time Frame: as for outcome 1
Population: The number analyzed reflects participants who experienced swelling at the specified location (axilla or supraclavicular) and the side relative to vaccine administration. For example, "Duration of LN swelling - Supraclavicular, Contralateral to Vaccine: 24 hours or less" for Dose 1 included 11 patients, as 11 of 61 reported swelling in the supraclavicular region contralateral to the side they received the vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated Breast Cancer Patients Dose 1 [mRNA vaccine - Moderna, Pfizer] | Vaccinated Breast Cancer Patients Dose 2 [mRNA vaccine - Moderna, Pfizer] | Vaccinated Breast Cancer Patients Booster [mRNA vaccine - Moderna, Pfizer] | Vaccinated Breast Cancer Patients Dose 1 [Non-mRNA vaccine - Johnson & Johnson] | Vaccinated Breast Cancer Patients Booster [Non-mRNA vaccine - Johnson & Johnson]
Number analyzed (Participants) | 61 | 80 | 53 | 4 | 1
Participants
  Duration of LN swelling - Supraclavicular, Contralateral to Vaccine: 24 hours or less: number analyzed (Participants) | 11 | 16 | 5 | 4 | 1
  Duration of LN swelling - Supraclavicular, Contralateral to Vaccine: 24 hours or less | 2 | 2 | 0 | 0 | 0
  Duration of LN swelling - Supraclavicular, Contralateral to Vaccine: 48 hours or less: number analyzed (Participants) | 11 | 16 | 5 | 4 | 1
  Duration of LN swelling - Supraclavicular, Contralateral to Vaccine: 48 hours or less | 3 | 0 | 1 | 0 | 0
  Duration of LN swelling - Supraclavicular, Contralateral to Vaccine: 1 week or less: number analyzed (Participants) | 11 | 16 | 5 | 4 | 1
  Duration of LN swelling - Supraclavicular, Contralateral to Vaccine: 1 week or less | 2 | 4 | 2 | 0 | 0
  Duration of LN swelling - Supraclavicular, Contralateral to Vaccine: 2 weeks or less: number analyzed (Participants) | 11 | 16 | 5 | 4 | 1
  Duration of LN swelling - Supraclavicular, Contralateral to Vaccine: 2 weeks or less | 0 | 0 | 0 | 0 | 0
  Duration of LN swelling - Supraclavicular, Contralateral to Vaccine: 3 weeks or less: number analyzed (Participants) | 11 | 16 | 5 | 4 | 1
  Duration of LN swelling - Supraclavicular, Contralateral to Vaccine: 3 weeks or less | 0 | 0 | 0 | 0 | 0
  Duration of LN swelling - Supraclavicular, Contralateral to Vaccine: 4 weeks or less: number analyzed (Participants) | 11 | 16 | 5 | 4 | 1
  Duration of LN swelling - Supraclavicular, Contralateral to Vaccine: 4 weeks or less | 0 | 2 | 0 | 0 | 0
  Duration of LN swelling-Supraclavicular, Contralateral to Vaccine: > than 4 weeks/still experiencing: number analyzed (Participants) | 11 | 16 | 5 | 4 | 1
  Duration of LN swelling-Supraclavicular, Contralateral to Vaccine: > than 4 weeks/still experiencing | 2 | 4 | 2 | 0 | 0
  Duration of LN swelling - Supraclavicular, Contralateral to Vaccine: I don't know: number analyzed (Participants) | 11 | 16 | 5 | 4 | 1
  Duration of LN swelling - Supraclavicular, Contralateral to Vaccine: I don't know | 2 | 3 | 0 | 0 | 0
  Duration of LN swelling - Supraclavicular, Contralateral to Vaccine: Missing: number analyzed (Participants) | 11 | 16 | 5 | 4 | 1
  Duration of LN swelling - Supraclavicular, Contralateral to Vaccine: Missing | 0 | 1 | 0 | 0 | 0
  Duration of LN swelling - Supraclavicular, Ipsilateral to Vaccine: 24 hours or less: number analyzed (Participants) | 18 | 21 | 17 | 4 | 1
  Duration of LN swelling - Supraclavicular, Ipsilateral to Vaccine: 24 hours or less | 6 | 8 | 3 | 0 | 0
  Duration of LN swelling - Supraclavicular, Ipsilateral to Vaccine: 48 hours or less: number analyzed (Participants) | 18 | 21 | 17 | 4 | 1
  Duration of LN swelling - Supraclavicular, Ipsilateral to Vaccine: 48 hours or less | 6 | 2 | 2 | 0 | 0
  Duration of LN swelling - Supraclavicular, Ipsilateral to Vaccine: 1 week or less: number analyzed (Participants) | 18 | 21 | 17 | 4 | 1
  Duration of LN swelling - Supraclavicular, Ipsilateral to Vaccine: 1 week or less | 2 | 4 | 6 | 0 | 0
  Duration of LN swelling - Supraclavicular, Ipsilateral to Vaccine: 2 weeks or less: number analyzed (Participants) | 18 | 21 | 17 | 4 | 1
  Duration of LN swelling - Supraclavicular, Ipsilateral to Vaccine: 2 weeks or less | 0 | 0 | 1 | 0 | 0
  Duration of LN swelling - Supraclavicular, Ipsilateral to Vaccine: 3 weeks or less: number analyzed (Participants) | 18 | 21 | 17 | 4 | 1
  Duration of LN swelling - Supraclavicular, Ipsilateral to Vaccine: 3 weeks or less | 0 | 0 | 0 | 0 | 0
  Duration of LN swelling - Supraclavicular, Ipsilateral to Vaccine: 4 weeks or less: number analyzed (Participants) | 18 | 21 | 17 | 4 | 1
  Duration of LN swelling - Supraclavicular, Ipsilateral to Vaccine: 4 weeks or less | 0 | 1 | 0 | 0 | 0
  Duration of LN swelling - Supraclavicular, Ipsilateral to Vaccine: > than 4 weeks/still experiencing: number analyzed (Participants) | 18 | 21 | 17 | 4 | 1
  Duration of LN swelling - Supraclavicular, Ipsilateral to Vaccine: > than 4 weeks/still experiencing | 3 | 4 | 4 | 0 | 0
  Duration of LN swelling - Supraclavicular, Ipsilateral to Vaccine: I don't know: number analyzed (Participants) | 18 | 21 | 17 | 4 | 1
  Duration of LN swelling - Supraclavicular, Ipsilateral to Vaccine: I don't know | 1 | 2 | 1 | 1 | 0
  Duration of LN swelling - Axilla, Ipsilateral to Vaccine: 24 hours or less: number analyzed (Participants) | 33 | 50 | 38 | 4 | 1
  Duration of LN swelling - Axilla, Ipsilateral to Vaccine: 24 hours or less | 2 | 6 | 2 | 0 | 0
  Duration of LN swelling - Axilla, Ipsilateral to Vaccine: 48 hours or less: number analyzed (Participants) | 33 | 50 | 38 | 4 | 1
  Duration of LN swelling - Axilla, Ipsilateral to Vaccine: 48 hours or less | 9 | 7 | 4 | 0 | 0
  Duration of LN swelling - Axilla, Ipsilateral to Vaccine: 1 week or less: number analyzed (Participants) | 33 | 50 | 38 | 4 | 1
  Duration of LN swelling - Axilla, Ipsilateral to Vaccine: 1 week or less | 10 | 17 | 19 | 0 | 0
  Duration of LN swelling - Axilla, Ipsilateral to Vaccine: 2 weeks or less: number analyzed (Participants) | 33 | 50 | 38 | 4 | 1
  Duration of LN swelling - Axilla, Ipsilateral to Vaccine: 2 weeks or less | 3 | 0 | 1 | 0 | 0
  Duration of LN swelling - Axilla, Ipsilateral to Vaccine: 3 weeks or less: number analyzed (Participants) | 33 | 50 | 38 | 4 | 1
  Duration of LN swelling - Axilla, Ipsilateral to Vaccine: 3 weeks or less | 1 | 2 | 3 | 0 | 0
  Duration of LN swelling - Axilla, Ipsilateral to Vaccine: 4 weeks or less: number analyzed (Participants) | 33 | 50 | 38 | 4 | 1
  Duration of LN swelling - Axilla, Ipsilateral to Vaccine: 4 weeks or less | 1 | 2 | 3 | 0 | 0
  Duration of LN swelling - Axilla, Ipsilateral to Vaccine: More than 4 weeks/still experiencing: number analyzed (Participants) | 33 | 50 | 38 | 4 | 1
  Duration of LN swelling - Axilla, Ipsilateral to Vaccine: More than 4 weeks/still experiencing | 3 | 10 | 3 | 1 | 0
  Duration of LN swelling - Axilla, Ipsilateral to Vaccine: I don't know: number analyzed (Participants) | 33 | 50 | 38 | 4 | 1
  Duration of LN swelling - Axilla, Ipsilateral to Vaccine: I don't know | 4 | 5 | 3 | 2 | 0
  Duration of LN swelling - Axilla, Ipsilateral to Vaccine: Missing: number analyzed (Participants) | 33 | 50 | 38 | 4 | 1
  Duration of LN swelling - Axilla, Ipsilateral to Vaccine: Missing | 0 | 1 | 0 | 0 | 0
  Duration of LN swelling - Axilla, Contralateral to Vaccine: 24 hours or less: number analyzed (Participants) | 28 | 36 | 13 | 4 | 1
  Duration of LN swelling - Axilla, Contralateral to Vaccine: 24 hours or less | 2 | 2 | 0 | 0 | 0
  Duration of LN swelling - Axilla, Contralateral to Vaccine: 48 hours or less: number analyzed (Participants) | 28 | 36 | 13 | 4 | 1
  Duration of LN swelling - Axilla, Contralateral to Vaccine: 48 hours or less | 2 | 2 | 2 | 0 | 0
  Duration of LN swelling - Axilla, Contralateral to Vaccine: 1 week or less: number analyzed (Participants) | 28 | 36 | 13 | 4 | 1
  Duration of LN swelling - Axilla, Contralateral to Vaccine: 1 week or less | 6 | 9 | 5 | 0 | 0
  Duration of LN swelling - Axilla, Contralateral to Vaccine: 2 weeks or less: number analyzed (Participants) | 28 | 36 | 13 | 4 | 1
  Duration of LN swelling - Axilla, Contralateral to Vaccine: 2 weeks or less | 3 | 3 | 0 | 0 | 0
  Duration of LN swelling - Axilla, Contralateral to Vaccine: 3 weeks or less: number analyzed (Participants) | 28 | 36 | 13 | 4 | 1
  Duration of LN swelling - Axilla, Contralateral to Vaccine: 3 weeks or less | 1 | 2 | 0 | 0 | 0
  Duration of LN swelling - Axilla, Contralateral to Vaccine: 4 weeks or less: number analyzed (Participants) | 28 | 36 | 13 | 4 | 1
  Duration of LN swelling - Axilla, Contralateral to Vaccine: 4 weeks or less | 3 | 4 | 1 | 0 | 0
  Duration of LN swelling - Axilla, Contralateral to Vaccine: More than 4 weeks/still experiencing: number analyzed (Participants) | 28 | 36 | 13 | 4 | 1
  Duration of LN swelling - Axilla, Contralateral to Vaccine: More than 4 weeks/still experiencing | 8 | 13 | 3 | 0 | 1
  Duration of LN swelling - Axilla, Contralateral to Vaccine: I don't know: number analyzed (Participants) | 28 | 36 | 13 | 4 | 1
  Duration of LN swelling - Axilla, Contralateral to Vaccine: I don't know | 3 | 1 | 2 | 0 | 0

4. Primary Outcome: Reported Side Effects of the mRNA and Non-mRNA Vaccines
Description: Due to the inherent activity of mRNA vaccines and the immune system, as well as the role of the lymph nodes in breast cancer (BC) and in breast cancer-related lymphedema (BCRL), this study analyzed the side effect profile in patients treated for BC and who received up to three doses of the COVID-19 vaccinations [Moderna, Pfizer]. A separate analysis is presented on results from participants who received the Johnson & Johnson (J&J) vaccine as lymph node swelling is not a listed side effect of this non-mRNA vaccine and only a small proportion of the population received this vaccine.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- [mRNA vaccine Dose 1- Moderna, Pfizer] reported side effects; [mRNA vaccine Dose 2- Moderna, Pfizer] reported side effects; [mRNA vaccine Booster - Moderna, Pfizer] reported side effects; [non-mRNA vaccine Dose 1 - Johnson & Johnson] reported side effects; [non-mRNA vaccine Booster - Johnson & Johnson] reported side effects: Patients who enroll in the trial and decided to get the COVID-19 vaccine will complete surveys to indicate their experiences, side effects, location of vaccination (i.e. right arm, left arm, or leg). This information will be analyzed in conjunction with their breast cancer treatment history and lymphedema measurements.
  Participants were separated into two different cohorts for analysis, Cohort 1 being those who received an mRNA vaccine for their primary vaccination series (two doses of Moderna or Pfizer) and Cohort 2 being those who received a non-mRNA vaccination for their primary vaccination series (one dose of Johnson & Johnson).
Arm/Group | [mRNA vaccine Dose 1- Moderna, Pfizer] reported side effects | [mRNA vaccine Dose 2- Moderna, Pfizer] reported side effects | [mRNA vaccine Booster - Moderna, Pfizer] reported side effects | [non-mRNA vaccine Dose 1 - Johnson & Johnson] reported side effects | [non-mRNA vaccine Booster - Johnson & Johnson] reported side effects
Number analyzed (Participants) | 621 | 621 | 469 | 49 | 34
Participants
  Symptom: Injection Site Soreness | 472 | 473 | 328 | 31 | 19
  Symptom: Fatigue | 265 | 368 | 208 | 21 | 10
  Symptom: Generalized Muscle Soreness | 143 | 198 | 115 | 9 | 5
  Symptom: Headache | 114 | 201 | 101 | 15 | 8
  Symptom: Chills | 59 | 147 | 90 | 10 | 5
  Symptom: Joint Pain | 58 | 108 | 59 | 8 | 4
  Symptom: Fever | 31 | 104 | 52 | 7 | 5
  Symptom: Injection Site Swelling | 84 | 119 | 63 | 5 | 2
  Symptom: Arm Heaviness | 60 | 59 | 30 | 2 | 2
  Symptom: Arm Swelling | 16 | 27 | 17 | 1 | 1
  Symptom: Vomiting | 4 | 7 | 6 | 0 | 1
  Symptom: Arm numbness | 13 | 12 | 8 | 0 | 0
  Symptom: Bell's Palsy | 0 | 0 | 0 | 0 | 0
  Symptom: Other | 27 | 34 | 27 | 1 | 0
  Symptom: None | 89 | 75 | 72 | 13 | 10

5. Primary Outcome: Duration of Side Effects of mRNA and Non-mRNA Vaccines
Description: Due to the inherent activity of mRNA vaccines and the immune system, as well as the role of the lymph nodes in breast cancer (BC) and in breast cancer-related lymphedema (BCRL), this study analyzed the side effect profile in patients treated for BC and who received up to three doses of the COVID-19 vaccinations [Moderna, Pfizer]. A separate analysis is presented on results from participants who received the Johnson & Johnson (J&J) vaccine as lymph node swelling is not a listed side effect of this non-mRNA vaccine and only a small proportion of the population received this vaccine.
  This outcome analyzes the duration of side effects associated with each dose of the vaccine.
Time Frame: as for outcome 1
Population: Participants are represented in multiple rows for the duration of separate side effects, so they can be accounted for in more than one row. The discrepancy for the "[mRNA vaccine Dose 1 - Moderna, Pfizer] reported side effects" Arm/Group is due to three participants who did not respond to the side effects question for Dose 1, resulting in a total of 529 responses out of 532 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | [mRNA vaccine Dose 1- Moderna, Pfizer] reported side effects | [mRNA vaccine Dose 2- Moderna, Pfizer] reported side effects | [mRNA vaccine Booster - Moderna, Pfizer] reported side effects | [non-mRNA vaccine Dose 1 - Johnson & Johnson] reported side effects | [non-mRNA vaccine Booster - Johnson & Johnson] reported side effects
Number analyzed (Participants) | 529 | 556 | 397 | 36 | 24
Participants
  24 hours or less | 218 | 215 | 175 | 16 | 12
  48 hours or less | 205 | 202 | 144 | 13 | 10
  1 week or less | 67 | 92 | 76 | 3 | 0
  2 weeks or less | 9 | 8 | 8 | 1 | 2
  3 weeks or less | 3 | 4 | 3 | 0 | 0
  4 weeks or less | 5 | 11 | 4 | 0 | 0
  More than 4 weeks/still experiencing | 14 | 29 | 10 | 1 | 1
  I don't know | 8 | 8 | 5 | 2 | 0

ADVERSE EVENTS:
Time Frame: This was a survey study of patients with breast surgery for breast cancer. Participants replied to the online survey up to 361.5 months post their breast surgery (median 69.0 months). This was the study's reported timeframe in the published manuscript. This was a non-interventional cross-sectional survey study. There were no adverse events reported as there was no study intervention.
Description: This was a non-interventional cross-sectional survey study. There were no adverse events reported as there was no study intervention.
Groups:
- Vaccinated Breast Cancer Patients [mRNA Vaccine Dose 1- Moderna, Pfizer]: Patients who enroll in the trial and decided to get the COVID-19 vaccine will complete surveys to indicate their experiences, side effects, location of vaccination (i.e. right arm, left arm, or leg). This information will be analyzed in conjunction with their breast cancer treatment history and lymphedema measurements.
  Participants were separated into two different cohorts for analysis, Cohort 1 being those who received an mRNA vaccine for their primary vaccination series (two doses of Moderna or Pfizer) and Cohort 2 being those who received a non-mRNA vaccination for their primary vaccination series (one dose of Johnson & Johnson).
  Side effects were reported separately for each vaccine dose and booster. The data presented here represent Dose 1 of the mRNA vaccine cohort.
  Survey: Patients in all groups will complete surveys about their experience with the vaccination and any side effects they may have experienced.
- Vaccinated Breast Cancer Patients [mRNA Vaccine Dose 2- Moderna, Pfizer]: Patients who enroll in the trial and decided to get the COVID-19 vaccine will complete surveys to indicate their experiences, side effects, location of vaccination (i.e. right arm, left arm, or leg). This information will be analyzed in conjunction with their breast cancer treatment history and lymphedema measurements.
  Participants were separated into two different cohorts for analysis, Cohort 1 being those who received an mRNA vaccine for their primary vaccination series (two doses of Moderna or Pfizer) and Cohort 2 being those who received a non-mRNA vaccination for their primary vaccination series (one dose of Johnson & Johnson).
  Side effects were reported separately for each vaccine dose and booster. The data presented here represent Dose 2 of the mRNA vaccine cohort.
  Survey: Patients in all groups will complete surveys about their experience with the vaccination and any side effects they may have experienced.
- Vaccinated Breast Cancer Patients [mRNA Vaccine Booster - Moderna, Pfizer]: Patients who enroll in the trial and decided to get the COVID-19 vaccine will complete surveys to indicate their experiences, side effects, location of vaccination (i.e. right arm, left arm, or leg). This information will be analyzed in conjunction with their breast cancer treatment history and lymphedema measurements.
  Participants were separated into two different cohorts for analysis, Cohort 1 being those who received an mRNA vaccine for their primary vaccination series (two doses of Moderna or Pfizer) and Cohort 2 being those who received a non-mRNA vaccination for their primary vaccination series (one dose of Johnson & Johnson).
  Side effects were reported separately for each vaccine dose and booster. The data presented here represents patients who received the mRNA vaccine booster.
  Survey: Patients in all groups will complete surveys about their experience with the vaccination and any side effects they may have experienced.
- Vaccinated Breast Cancer Patients [Non-mRNA Vaccine Dose 1 - Johnson & Johnson]: Patients who enroll in the trial and decided to get the COVID-19 vaccine will complete surveys to indicate their experiences, side effects, location of vaccination (i.e. right arm, left arm, or leg). This information will be analyzed in conjunction with their breast cancer treatment history and lymphedema measurements.
  Participants were separated into two different cohorts for analysis, Cohort 1 being those who received an mRNA vaccine for their primary vaccination series (two doses of Moderna or Pfizer) and Cohort 2 being those who received a non-mRNA vaccination for their primary vaccination series (one dose of Johnson & Johnson).
  Side effects were reported separately for each vaccine dose and booster. The data presented here represents the non-mRNA vaccine cohort.
  Survey: Patients in all groups will complete surveys about their experience with the vaccination and any side effects they may have experienced.
- Vaccinated Breast Cancer Patients [Non-mRNA Vaccine Booster - Johnson & Johnson]: Patients who enroll in the trial and decided to get the COVID-19 vaccine will complete surveys to indicate their experiences, side effects, location of vaccination (i.e. right arm, left arm, or leg). This information will be analyzed in conjunction with their breast cancer treatment history and lymphedema measurements.
  Participants were separated into two different cohorts for analysis, Cohort 1 being those who received an mRNA vaccine for their primary vaccination series (two doses of Moderna or Pfizer) and Cohort 2 being those who received a non-mRNA vaccination for their primary vaccination series (one dose of Johnson & Johnson).
  Side effects were reported separately for each vaccine dose and booster. The data presented here represents patients who received the non-mRNA vaccine booster.
  Survey: Patients in all groups will complete surveys about their experience with the vaccination and any side effects they may have experienced.
Arm/Group | Vaccinated Breast Cancer Patients [mRNA Vaccine Dose 1- Moderna, Pfizer] | Vaccinated Breast Cancer Patients [mRNA Vaccine Dose 2- Moderna, Pfizer] | Vaccinated Breast Cancer Patients [mRNA Vaccine Booster - Moderna, Pfizer] | Vaccinated Breast Cancer Patients [Non-mRNA Vaccine Dose 1 - Johnson & Johnson] | Vaccinated Breast Cancer Patients [Non-mRNA Vaccine Booster - Johnson & Johnson]
All-Cause Mortality (participants affected / at risk) | 9/621 | 3/621 | 0/469 | 0/49 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/621 | 0/621 | 0/469 | 0/49 | 0/34
Other Adverse Events (participants affected / at risk) | 532/621 | 546/621 | 397/469 | 36/49 | 24/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccinated Breast Cancer Patients [mRNA Vaccine Dose 1- Moderna, Pfizer] (N=621) | Vaccinated Breast Cancer Patients [mRNA Vaccine Dose 2- Moderna, Pfizer] (N=621) | Vaccinated Breast Cancer Patients [mRNA Vaccine Booster - Moderna, Pfizer] (N=469) | Vaccinated Breast Cancer Patients [Non-mRNA Vaccine Dose 1 - Johnson & Johnson] (N=49) | Vaccinated Breast Cancer Patients [Non-mRNA Vaccine Booster - Johnson & Johnson] (N=34)
Injection Site Soreness (General disorders) | 472 | 473 | 328 | 31 | 19
Injection site swelling (Skin and subcutaneous tissue disorders) | 84 | 119 | 63 | 5 | 2
Injection site redness (Skin and subcutaneous tissue disorders) | 76 | 85 | 52 | 4 | 1
Arm swelling (Skin and subcutaneous tissue disorders) | 16 | 27 | 17 | 1 | 1
Arm numbness (Skin and subcutaneous tissue disorders) | 13 | 12 | 8 | 0 | 0
Arm heaviness (Musculoskeletal and connective tissue disorders) | 60 | 59 | 30 | 2 | 2
Generalized muscle soreness (Musculoskeletal and connective tissue disorders) | 143 | 198 | 115 | 9 | 5
Fatigue (General disorders) | 265 | 368 | 208 | 21 | 10
Headache (General disorders) | 114 | 201 | 101 | 15 | 8
Joint Pain (Musculoskeletal and connective tissue disorders) | 58 | 108 | 59 | 8 | 4
Chills (General disorders) | 59 | 147 | 90 | 10 | 5
Nausea (Gastrointestinal disorders) | 33 | 53 | 25 | 4 | 4
Vomiting (Gastrointestinal disorders) | 4 | 7 | 6 | 0 | 1
Fever (General disorders) | 31 | 104 | 52 | 7 | 5
Bell's Palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0
LN Swelling (Blood and lymphatic system disorders) | 61 | 80 | 53 | 4 | 1

LIMITATIONS AND CAVEATS:
It is difficult to determine the exact response rate as surveys were sent when many patients hadn't yet received the vaccine; recall bias may have played a role.

Questions regarding LN swelling relied on self-report.

The surveys do not include questions regarding the severity of the side effects reported; therefore, conclusions about severity cannot be drawn.

Methodological limitations prevent statistical comparisons with studies of the general population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT04872738/Prot_SAP_000.pdf